CLINICAL TRIAL: NCT01079910
Title: Clinical Efficacy of an Experimental Toothpaste
Brief Title: To Investigate the Clinical Efficacy of an Experimental Toothpaste
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: T3450803
Record Dates: First submitted 2010-02-18; First posted 2010-03-03 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Gingivitis
Keywords: Plaque; Toothpaste; Gingivitis
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid | interventions — Fluorides; Silicon Dioxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental toothpaste (Experimental): 0.1% isopropylmethylphenol and 1150ppm fluoride
  Interventions: Drug: isopropylmethylphenol and Fluoride
- Marketed toothpaste (Other): NaF/Silica toothpaste containing 1150ppm fluoride
  Interventions: Drug: Fluoride and Silica

INTERVENTIONS:
Drug: isopropylmethylphenol and Fluoride — 0.1% isopropylmethylphenol and 1150ppm fluoride
  Arms: Experimental toothpaste
Drug: Fluoride and Silica — NaF/Silica toothpaste containing 1150ppm fluoride
  Arms: Marketed toothpaste

SUMMARY:
The objective of this study is to evaluate the effect of an experimental toothpaste on maintaining gingival health over a 24 week period measured through modified gingival index, bleeding, plaque, and plaque bacteria. Prior to commencing study treatment, subjects will undergo a dental prophylaxis followed by a 2 week period of oral hygiene instruction and weekly professional tooth cleaning to bring the subjects to their optimum gingival health prior to commencing study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 years and older
* A minimum of 20 permanent gradable teeth
* For baseline eligibility, subjects must have a minimum Modified Gingival Index score of 1.5-2.3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12-09 (Estimated); Primary Completion 2009-12-10 (Estimated); Study Completion 2009-12-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Modified Gingival Index at 24 weeks | baseline to 24 weeks
Change from baseline Bleeding Index at 24 weeks | baseline to 24 weeks

SECONDARY OUTCOMES:
Change from baseline Modified Gingival Index at weeks 6 & 12 | baseline to week 12
Change from baseline Bleeding Index at weeks 6 & 12 | baseline to week 12
Change from baseline Plaque Index at weeks 6, 12 & 24 | baseline to week 24
Change from baseline plaque bacteria at weeks 12 & 24 | baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline